CLINICAL TRIAL: NCT05658523
Title: A Randomised Controlled Trial to Assess the Immunogenicity, Safety and Reactogenicity of a Bivalent mRNA Moderna COVID-19 Vaccine or a Protein-based Novavax COVID-19 Vaccine Given as a Fourth Dose in Healthy Adults in Australia
Brief Title: COVID-19 Booster Study in Healthy Adults in Australia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other); The Peter Doherty Institute for Infection and Immunity (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 91108
Record Dates: First submitted 2022-12-19; First posted 2022-12-20 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: Booster dose Moderna and Novavax; control group; monovalent, bivalent
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273; mRNA-1273.214 COVID-19 vaccine; NVX-CoV2373 adjuvated lipid nanoparticle

STUDY DESIGN:
Intervention Model Description: Study participants who have previously received 3 COVID-19 vaccines will be either randomised into one of two vaccine groups or be part of a self-selected control group. Randomised participants will receive a standard dose of either the bivalent Moderna or the protein-based Novavax vaccine. 200 non-randomised participants will be part of a control group and will not receive any COVID-19 vaccine.
Who Masked: Participant, Investigator
Masking Description: The participants and those evaluating reactogenicity will be blinded to the vaccine allocation for the first 7 days following vaccination. After that, both clinical investigators and participants will be aware of their investigational product. Laboratory staff will remain blinded to the investigational product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Bivalent Moderna (mRNA-1273.214) (Active Comparator): Participants who have received three doses of COVID-19 vaccine, with the last dose at least 6 months prior to the study, will receive a booster dose of bivalent mRNA Moderna COVID-19 vaccine (mRNA-1273.214)
  The mRNA-1273.214 encodes the prefusion stabilized S protein of SARS-CoV-2 formulated in RNA-lipid nanoparticles composed of 4 lipids and 1-monomethoxypolyethyleneglycol-2, 3-dimyristylglycerol with polyethylene glycol. 25μg of each mRNA sequence that encode the prefusion stabilized spike glycoproteins of the ancestral SARS-CoV-2 (Wuhan-Hu-1) and the Omicron variant (B.1.1.529 [BA.1]).
  Interventions: Biological: Bivalent Moderna
- Novavax (Active Comparator): Participants who have received three doses of COVID-19 vaccine, with the last dose at least 6 months prior to the study, will receive a booster dose of Novavax COVID-19 protein subunit vaccine.
  Novavax contains 5μg of SARS-CoV-2 spike protein and is adjuvanted with Matrix-M. Adjuvant Matrix-M contains, per 0.5 mL dose: Quillaja saponaria saponins fraction A (42.5 micrograms) and Quillaja saponaria saponins fraction C (7.5 micrograms).
  Interventions: Biological: Novavax
- Control group- no vaccine (No Intervention): Participants who have received three doses of COVID-19 vaccine, with the last dose at least 6 months prior to the study, will be recruited but will not receive any COVID-19 vaccine.

INTERVENTIONS:
Biological: Bivalent Moderna — A single standard dose of the bivalent Moderna (mRNA-1273.214) COVID-19 vaccine containing equal amounts of mRNAs (25μg of each mRNA sequence) that encode the prefusion stabilized spike glycoproteins of the ancestral SARS-CoV-2 (Wuhan-Hu-1) and the Omicron variant (B.1.1.529 [BA.1]) with mRNAs encapsulated in lipid nanoparticles, will be administered on day 0 of the study.
  Other Names: mRNA-1273.214
  Arms: Bivalent Moderna (mRNA-1273.214)
Biological: Novavax — A single dose of Novavax contains 5μg of SARS-CoV-2 spike protein and is adjuvanted with Matrix-M. Adjuvant Matrix-M contains, per 0.5 mL dose: Quillaja saponaria saponins fraction A (42.5 micrograms) and Quillaja saponaria saponins fraction C (7.5 micrograms), will be administered on day 0 of the study.
  Arms: Novavax

SUMMARY:
This is a double-blinded, randomised study to determine the safety, reactogenicity, and immunogenicity of a bivalent mRNA Moderna COVID-19 vaccine or a protein-based Novavax COVID-19 vaccine given as a fourth dose in healthy adults in Australia.

DETAILED DESCRIPTION:
This is a blinded, two-arm randomised study to determine the safety, reactogenicity and immunogenicity of a fourth dose of SARS-CoV-2 vaccines in Australia in adults 18 years or older who have received their third dose of COVID-19 vaccine at least six months previously. Participants will be randomised to receive either bivalent Moderna (mRNA-1273.214) or Novavax. A separate non-randomised control arm (no vaccine given), frequency matched by age to the vaccine groups will also be enrolled for comparison. A total of 200 participants per group will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Have received three doses of COVID-19 vaccines at least 6 months earlier.
2. No confirmed SARS-CoV-2 infection on PCR or RAT within the last 3 months.
3. Willing and able to give written informed consent.
4. Aged 18 years or above.
5. Willing to complete the follow-up requirements of the study.

Exclusion Criteria:

1. Currently receiving immunosuppressive medication or anti-cancer chemotherapy.
2. Known HIV infection.
3. Congenital immune deficiency syndrome.
4. Received immunoglobulin or other blood products in the three months prior to potential study booster vaccination.
5. Study staff and their relatives.
6. Have a history of a severe allergic reaction to any COVID-19 vaccines or have a medical exemption to receiving further COVID-19 vaccines.
7. Cannot read or understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-10-13 (Actual); Study Completion 2026-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Mulholland, MD/Prof, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Royal Children's Hospital, Murdoch Children's Research Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share de-identified data to ethically approved studies in cases where participants have indicated on the consent form that they consent to the use of their data and where consistent with terms of collaboration agreements.
Supporting Information: Study Protocol, ICF
Time Frame: Individual participant data (IPD) sharing plans in development
Access Criteria: In development

REFERENCES:
- See also: Coalition for Epidemic Preparedness Innovations (CEPI). Priority List of Adverse Events of Special Interest: COVID-19 2020 [Available from: — https://media.tghn.org/articles/COVID-19_AESIs_SPEAC_V1.1_5Mar2020.pdf
- See also: World Health Organization. Interim statement on the use of additional booster doses of Emergency Use Listed mRNA vaccines against COVID-19 2022 — https://www.who.int/news/item/17-05-2022-interim-statement-on-the-use-of-additional-booster-doses-of-emergency-use-listed-mrna-vaccines-against-covid-19
- See also: US Food and Drug Administration (FDA). Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials 2007 — https://www.fda.gov/media/73679/download
- See also: International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use. Addendum on Estimands and Sensitivity Analysis in Clinical Trials to the Guideline on Statistical Principles for Clinical Trials 2019 — https://database.ich.org/sites/default/files/E9-R1_Step4_Guideline_2019_1203.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Bivalent Moderna (mRNA-1273.214): Participants who have received three doses of COVID-19 vaccine, with the last dose at least 6 months prior to the study, will receive a booster dose of bivalent mRNA Moderna COVID-19 vaccine (mRNA-1273.214)
  The mRNA-1273.214 encodes the prefusion stabilized S protein of SARS-CoV-2 formulated in RNA-lipid nanoparticles composed of 4 lipids and 1-monomethoxypolyethyleneglycol-2, 3-dimyristylglycerol with polyethylene glycol. 25μg of each mRNA sequence that encode the prefusion stabilized spike glycoproteins of the ancestral SARS-CoV-2 (Wuhan-Hu-1) and the Omicron variant (B.1.1.529 [BA.1]).
  Bivalent Moderna: A single standard dose of the bivalent Moderna (mRNA-1273.214) COVID-19 vaccine containing equal amounts of mRNAs (25μg of each mRNA sequence) that encode the prefusion stabilized spike glycoproteins of the ancestral SARS-CoV-2 (Wuhan-Hu-1) and the Omicron variant (B.1.1.529 [BA.1]) with mRNAs encapsulated in lipid nanoparticles, will be administered on day 0 of the study.
- Novavax: Participants who have received three doses of COVID-19 vaccine, with the last dose at least 6 months prior to the study, will receive a booster dose of Novavax COVID-19 protein subunit vaccine.
  Novavax contains 5μg of SARS-CoV-2 spike protein and is adjuvanted with Matrix-M. Adjuvant Matrix-M contains, per 0.5 mL dose: Quillaja saponaria saponins fraction A (42.5 micrograms) and Quillaja saponaria saponins fraction C (7.5 micrograms).
  Novavax: A single dose of Novavax contains 5μg of SARS-CoV-2 spike protein and is adjuvanted with Matrix-M. Adjuvant Matrix-M contains, per 0.5 mL dose: Quillaja saponaria saponins fraction A (42.5 micrograms) and Quillaja saponaria saponins fraction C (7.5 micrograms), will be administered on day 0 of the study.
Period: Baseline
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Control Group- no Vaccine
Started | 177 | 176 | 143
Completed | 176 (One participant did not have blood taken) | 176 | 143
Not Completed | 1 | 0 | 0
Not completed — No blood draw | 1 | 0 | 0
Period: 28 Days
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Control Group- no Vaccine
Started | 177 | 176 | 143
Completed | 175 | 171 | 143
Not Completed | 2 | 5 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Visit missed | 0 | 4 | 0
Period: 6 Months
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Control Group- no Vaccine
Started | 175 | 175 | 143
Completed | 168 | 158 | 136
Not Completed | 7 | 17 | 7
Not completed — Lost to Follow-up | 1 | 7 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 4
Not completed — Visit missed | 5 | 7 | 0
Not completed — No blood draw | 0 | 0 | 1
Period: 12 Months
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Control Group- no Vaccine
Started | 173 | 165 | 137
Completed | 163 | 147 | 124
Not Completed | 10 | 18 | 13
Not completed — Lost to Follow-up | 2 | 6 | 3
Not completed — Withdrawal by Subject | 4 | 4 | 2
Not completed — Visit missed | 4 | 8 | 8
Period: 18 Months
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Control Group- no Vaccine
Started | 167 | 155 | 132
Completed | 133 | 124 | 108
Not Completed | 34 | 31 | 24
Not completed — Lost to Follow-up | 5 | 8 | 2
Not completed — Withdrawal by Subject | 17 | 9 | 16
Not completed — Visit missed | 12 | 14 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Control Group- no Vaccine | Total
Number analyzed (Participants) | 177 | 176 | 143 | 496
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age is recorded as a continuous variable in years at the time of booster vaccination. Values are derived from date of birth and visit date, and summarised using mean, standard deviation, median, and range to describe the baseline age distribution of participants
  years | 30 [26 to 42] | 31 [25 to 43] | 39 [29 to 51] | 32 [26 to 47]
Age, Customized [Count of Participants; unit: Participants] — Age is summarised in two strata (≥18 to <50 and ≥50 years) because randomisation was stratified by these groups. Age in completed years was derived from date of birth and visit date.
  Participants
    ≥18 to <50 years | 150 | 150 | 101 | 401
    ≥50 years | 27 | 26 | 42 | 95
Sex: Female, Male [Count of Participants; unit: Participants] — Sex was recorded as male or female based on participant self-report at enrolment.
  Participants
    Female | 116 | 128 | 114 | 358
    Male | 61 | 48 | 29 | 138
Region of Enrollment [Count of Participants; unit: Participants] — Region of enrolment reflects the geographic location where participants entered the study. All participants were enrolled in Melbourne, Victoria, Australia.
  Participants
    Australia | 177 | 176 | 143 | 496
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Body mass index (BMI) was calculated as weight in kilograms divided by height in metres squared (kg/m^2). BMI is presented as a continuous variable and summarised using the median and interquartile range Population: One participant is missing a weight measurement, as they declined the assessment.
  kg/m^2
    number analyzed (Participants) | 176 | 176 | 143 | 495
    (all) | 24.7 [21.2 to 27.2] | 24.8 [21.7 to 28.4] | 24.2 [21.7 to 27.5] | 24.5 [21.5 to 27.7]
Number of times tested positive for SARS-CoV-2 [Count of Participants; unit: Participants] — Participants were asked whether they had ever tested positive for SARS-CoV-2 before enrolment. If yes, they were then asked how many times they had tested positive in separate instances of infection.
  Participants
    0 prior positive SARS-CoV-2 tests | 37 | 30 | 42 | 109
    1 prior positive SARS-CoV-2 tests | 109 | 113 | 69 | 291
    2 prior positive SARS-CoV-2 tests | 26 | 28 | 28 | 82
    3 prior positive SARS-CoV-2 tests | 5 | 4 | 4 | 13
    4 prior positive SARS-CoV-2 tests | 0 | 1 | 0 | 1
Comorbidities [Count of Participants; unit: Participants] — Population: One participant is missing a weight measurement, as they declined the assessment. One participant is missing an observation for history of anaphylaxis. Therefore, there is an observation missing for the comorbidity of obesity (BMI ≥30 kg/m^2) and for history of anaphylaxis
  Participants
    Diabetes mellitus | 4 | 4 | 3 | 11
    Gestational diabetes | 0 | 1 | 1 | 2
    Obesity (BMI ≥30 kg/m^2): number analyzed (Participants) | 176 | 176 | 143 | 495
    Obesity (BMI ≥30 kg/m^2) | 27 | 33 | 21 | 81
    Cardiovascular disease | 1 | 3 | 1 | 5
    Hypertension | 8 | 9 | 8 | 25
    Cancer | 2 | 0 | 0 | 2
    Chronic obstructive pulmonary disease | 0 | 0 | 0 | 0
    Chronic kidney disease | 1 | 0 | 1 | 2
    Chronic liver disease | 1 | 0 | 2 | 3
    History of anaphylaxis: number analyzed (Participants) | 176 | 176 | 143 | 495
    History of anaphylaxis | 3 | 2 | 2 | 7
    Neurological disease | 1 | 2 | 1 | 4
    On anticoagulant therapy | 2 | 2 | 4 | 8
    Cigarette user | 5 | 7 | 0 | 12
    Pregnant at time of enrolment | 1 | 1 | 1 | 3
    Asthma | 25 | 28 | 19 | 72
    History of mastocytosis | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was self-reported and categorised according to U.S. OMB standards required by ClinicalTrials.gov. Participants identifying as Indigenous Australian were classified under 'American Indian or Alaska Native,' following ClinicalTrials.gov guidance for Indigenous populations.
  Participants
    American Indian or Alaska Native | 2 | 0 | 1 | 3
    Asian | 41 | 33 | 58 | 132
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 2 | 0 | 2
    White | 129 | 139 | 84 | 352
    More than one race | 3 | 0 | 0 | 3
    Unknown or Not Reported | 2 | 2 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was self-reported and categorised using the two U.S. OMB classifications required by ClinicalTrials.gov: 'Hispanic or Latino' and 'Not Hispanic or Latino.' Participants who selected 'Prefer not to say' were classified as 'Unknown/Not Reported.'
  Participants
    Hispanic or Latino | 0 | 2 | 1 | 3
    Not Hispanic or Latino | 175 | 172 | 142 | 489
    Unknown or Not Reported | 2 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: SARS-CoV-2 Specific Immunoglobulin (Ig)G Antibodies at 28-days Post Booster Vaccination
Description: Serum samples collected at 28-days post booster vaccination from the two intervention groups will be evaluated for SARS-CoV-2 specific IgG antibodies using the commercial Euroimmun S1 IgG ELISA. Data will be reported as binding antibody units/mL and presented as geometric mean concentration and 95% confidence intervals
Time Frame: 28-days post booster vaccination
Population: Moderna group:By day 28 1 participant was lost to follow-up and 1 had withdrawn Novavax: 4 people missed their visit for the day 28 blood draw and 1 was a withdrawal.
Measure: Geometric Mean (95% Confidence Interval); unit: binding antibody units (BAU/mL)
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax
Number analyzed (Participants) | 175 | 171
binding antibody units (BAU/mL) | 6792 [6191 to 7451] | 3179 [2854 to 3541]

2. Primary Outcome: Total Incidence of Solicited Reactions (Systemic and Local)
Description: Questionnaire to document solicited reactions is developed specifically for this study. Data will be reported as the proportion of participants who report by each intervention arm. Solicited reactions such as pain, tenderness, erythema/redness, induration/swelling, fever, nausea/vomiting, headache, fatigue/malaise, myalgia, arthralgia will be collected from the participants 7 days post-vaccination. Reactogenicity was graded on a 0-4 scale: Grade 0 = no symptom; Grade 1 = mild and does not interfere with activity; Grade 2 = moderate or requiring repeated non-narcotic analgesia; Grade 3 = severe, limiting or preventing daily activity; Grade 4 = potentially life-threatening, requiring ER visit or hospitalisation.
Time Frame: Total incidence of solicited reactions will be measured for 7 days post booster vaccination
Population: Solicited local and systemic reactions were collected for 7 days post-vaccination using a study-specific questionnaire. Outcomes are reported as both the number of participants in each arm and the percentage of participants in that arm experiencing reactions by severity grade. Reactions were graded on a 0-4 scale: Grade 0 = no symptom; Grade 1 = mild (does not interfere with activity); Grade 2 = moderate (may require non-narcotic analgesia); Grade 3 = severe (limits or prevents daily activity);
Measure: Count of Participants; unit: Participants
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax
Number analyzed (Participants) | 177 | 176
Participants
  Pain: Grade 0 no symptoms | 53 | 113
  Pain: Grade 1 (Mild) | 105 | 61
  Pain: Grade 2 Moderate | 19 | 2
  Pain: Grade 3 Severe | 0 | 0
  Pain: Grade 4 Potentially Life Threatening | 0 | 0
  Tenderness: Grade 0 no symptoms | 33 | 86
  Tenderness: Grade 1 (Mild) | 80 | 72
  Tenderness: Grade 2 Moderate | 60 | 16
  Tenderness: Grade 3 Severe | 4 | 2
  Tenderness: Grade 4 Potentially Life Threatening | 0 | 0
  Redness: Grade 0 no symptoms | 164 | 167
  Redness: Grade 1 (Mild) | 6 | 6
  Redness: Grade 2 Moderate | 5 | 3
  Redness: Grade 3 Severe | 1 | 0
  Redness: Grade 4 Potentially Life Threatening | 1 | 0
  Swelling: Grade 0 no symptoms | 157 | 172
  Swelling: Grade 1 (Mild) | 9 | 3
  Swelling: Grade 2 Moderate | 9 | 1
  Swelling: Grade 3 Severe | 1 | 0
  Swelling: Grade 4 Potentially Life Threatening | 1 | 0
  Hard: Grade 0 no symptoms | 157 | 171
  Hard: Grade 1 (Mild) | 14 | 4
  Hard: Grade 2 Moderate | 5 | 1
  Hard: Grade 3 Severe | 0 | 0
  Hard: Grade 4 Potentially Life Threatening | 1 | 0
  Axillary Lymphadenopathy: Grade 0 no symptoms | 149 | 162
  Axillary Lymphadenopathy: Grade 1 (Mild) | 21 | 13
  Axillary Lymphadenopathy: Grade 2 Moderate | 7 | 1
  Axillary Lymphadenopathy: Grade 3 Severe | 0 | 0
  Axillary Lymphadenopathy: Grade 4 Potentially Life Threatening | 0 | 0
  Warmth: Grade 0 no symptoms | 119 | 146
  Warmth: Grade 1 (Mild) | 55 | 29
  Warmth: Grade 2 Moderate | 3 | 1
  Warmth: Grade 3 Severe | 0 | 0
  Warmth: Grade 4 Potentially Life Threatening | 0 | 0
  Itch: Grade 0 no symptoms | 160 | 170
  Itch: Grade 1 (Mild) | 17 | 4
  Itch: Grade 2 Moderate | 0 | 2
  Itch: Grade 3 Severe | 0 | 0
  Itch: Grade 4 Potentially Life Threatening | 0 | 0
  Fever: Grade 0 no symptoms | 173 | 172
  Fever: Grade 1 (Mild) | 3 | 1
  Fever: Grade 2 Moderate | 1 | 0
  Fever: Grade 3 Severe | 0 | 2
  Fever: Grade 4 Potentially Life Threatening | 0 | 1
  Nausea: Grade 0 no symptoms | 147 | 159
  Nausea: Grade 1 (Mild) | 24 | 14
  Nausea: Grade 2 Moderate | 6 | 3
  Nausea: Grade 3 Severe | 0 | 0
  Nausea: Grade 4 Potentially Life Threatening | 0 | 0
  Vomiting: Grade 0 no symptoms | 173 | 174
  Vomiting: Grade 1 (Mild) | 4 | 2
  Vomiting: Grade 2 Moderate | 0 | 0
  Vomiting: Grade 3 Severe | 0 | 0
  Vomiting: Grade 4 Potentially Life Threatening | 0 | 0
  Diarrhoea: Grade 0 no symptoms | 163 | 163
  Diarrhoea: Grade 1 (Mild) | 12 | 11
  Diarrhoea: Grade 2 Moderate | 2 | 2
  Diarrhoea: Grade 3 Severe | 0 | 0
  Diarrhoea: Grade 4 Potentially Life Threatening | 0 | 0
  Headache: Grade 0 no symptoms | 81 | 127
  Headache: Grade 1 (Mild) | 61 | 40
  Headache: Grade 2 Moderate | 35 | 8
  Headache: Grade 3 Severe | 0 | 1
  Headache: Grade 4 Potentially Life Threatening | 0 | 0
  Fatigue/Malaise: Grade 0 no symptoms | 76 | 106
  Fatigue/Malaise: Grade 1 (Mild) | 54 | 44
  Fatigue/Malaise: Grade 2 Moderate | 42 | 22
  Fatigue/Malaise: Grade 3 Severe | 5 | 4
  Fatigue/Malaise: Grade 4 Potentially Life Threatening | 0 | 0
  Muscle pain: Grade 0 no symptoms | 94 | 140
  Muscle pain: Grade 1 (Mild) | 63 | 31
  Muscle pain: Grade 2 Moderate | 19 | 4
  Muscle pain: Grade 3 Severe | 1 | 1
  Muscle pain: Grade 4 Potentially Life Threatening | 0 | 0
  Joint pain: Grade 0 no symptoms | 128 | 157
  Joint pain: Grade 1 (Mild) | 36 | 16
  Joint pain: Grade 2 Moderate | 12 | 3
  Joint pain: Grade 3 Severe | 1 | 0
  Joint pain: Grade 4 Potentially Life Threatening | 0 | 0

3. Secondary Outcome: SARS-CoV-2 Specific IgG Antibodies at Baseline (Pre Booster), and 6,12 and 18 Months Post Booster Vaccination
Description: Serum samples collected at baseline (pre booster), 28 days, 6,12, 18, 24, and 30 months post booster vaccination from the two intervention groups and the control group will be evaluated for SARS-CoV-2 specific IgG antibodies using the commercial Euroimmun S1 IgG ELISA . Data will be reported as binding antibody units/mL and presented as geometric mean concentration and 95% confidence intervals
Time Frame: Baseline (pre booster), 6-months,12-months and 18-months post booster vaccination
Population: One person in the Moderna group didn't have a blood taken at baseline
Measure: Geometric Mean (95% Confidence Interval); unit: binding antibody units (BAU/mL)
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Control Group- no Vaccine
Number analyzed (Participants) | 176 | 176 | 143
binding antibody units (BAU/mL)
  Baseline anti-spike IgG GMC (95% CI) | 1418 [1222 to 1646] | 1434 [1257 to 1636] | 1182 [1003 to 1392]
  28 day anti-spike IgG GMC (95% CI) (Note, controls did not have blood taken at 28 days): number analyzed (Participants) | 175 | 171 | 0
  28 day anti-spike IgG GMC (95% CI) (Note, controls did not have blood taken at 28 days) | 6792 [6191 to 7452] | 3179 [2854 to 3541] |
  6 month anti-spike IgG GMC (95% CI): number analyzed (Participants) | 168 | 158 | 136
  6 month anti-spike IgG GMC (95% CI) | 2451 [2189 to 2745] | 1601 [1424 to 1801] | 1108 [931 to 1320]
  12 month anti-spike IgG GMC (95% CI): number analyzed (Participants) | 163 | 147 | 124
  12 month anti-spike IgG GMC (95% CI) | 2047 [1830 to 2289] | 1579 [1405 to 1775] | 1346 [1147 to 1580]
  18 month anti-spike IgG GMC (95% CI): number analyzed (Participants) | 133 | 123 | 108
  18 month anti-spike IgG GMC (95% CI) | 4059 [3415 to 4825] | 3103 [2616 to 3681] | 3186 [2560 to 3964]

4. Secondary Outcome: SARS-CoV-2 Specific Neutralising Antibodies Measured by Surrogate Virus Neutralization Test (sVNT)
Description: Neutralising antibody levels will be measured using the GenScript® cPass sVNT, which reports inhibition relative to a positive control. Results are expressed as concentrations (U/mL) and summarised as geometric mean concentrations (GMCs) with 95% CIs.
Time Frame: Baseline (pre booster), 28 days, 6,12, 18, 24, and 30 months post booster vaccination
Population: No Day 28 samples collected from control group as they did not receive any vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Control Group- no Vaccine
Number analyzed (Participants) | 176 | 176 | 143
U/mL
  Baseline Wuhan-Hu-1 SARS-CoV-2 sVNT U/mL GMC (95% CI) | 45745 [38942 to 53736] | 48790 [42339 to 56223] | 63280 [54378 to 73638]
  28 days Wuhan-Hu-1 SARS-CoV-2 sVNT U/mL GMC (95% CI): number analyzed (Participants) | 175 | 171 | 0
  28 days Wuhan-Hu-1 SARS-CoV-2 sVNT U/mL GMC (95% CI) | 224397 [204299 to 246472] | 96581 [86417 to 107941] |
  6 months Wuhan-Hu-1 SARS-CoV-2 sVNT U/mL GMC (95% CI): number analyzed (Participants) | 168 | 158 | 136
  6 months Wuhan-Hu-1 SARS-CoV-2 sVNT U/mL GMC (95% CI) | 92355 [81954 to 104077] | 63682 [56541 to 71724] | 48556 [41569 to 56716]
  12 months Wuhan-Hu-1 SARS-CoV-2 sVNT U/mL GMC (95% CI): number analyzed (Participants) | 163 | 147 | 124
  12 months Wuhan-Hu-1 SARS-CoV-2 sVNT U/mL GMC (95% CI) | 46494 [40992 to 52734] | 36869 [32362 to 41936] | 33932 [28989 to 39719]

5. Secondary Outcome: SARS-CoV-2 Specific Neutralising Antibodies at Baseline (Pre Booster), 28 Days and 6, 12 and 18 Months Post Booster Vaccination Measured by SARS-CoV-2 Microneutralisation Assay
Description: A subset of samples (20%) from all timepoints will be assessed using a SARS-CoV-2 microneutralisation assay to both the wild type (vaccine) strain and for two SARS-CoV-2 Variants of concern. Neutralizing antibody will be reported as endpoint titre.
Time Frame: Baseline (pre booster), 6,12 and 18-months post booster vaccination
Reporting Status: Not Posted

6. Secondary Outcome: Interferon Gamma (IFNγ) Concentrations in International Units (IU)/mL
Description: Interferon gamma (IFNγ) concentrations as a measurement of cellular immunity will be assessed on a subset (50%) of the participants from each group. QuantiFERON Human IFN-γ SARS-CoV-2 (Qiagen) will be used to stimulate IFN-γ production in whole blood and then IFN-γ production will be measured using Enzyme-Linked ImmunoSorbent Assay (ELISA). Data will be presented as geometric mean concentration (GMC) and 95% confidence intervals (CI).
Time Frame: Baseline (pre booster), Day 28, 6-months and 12-months post booster vaccination
Population: No Day 28 samples collected for Control group as no vaccine were given.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Control Group- no Vaccine
Number analyzed (Participants) | 89 | 89 | 73
IU/mL
  Baseline | 0.39 [0.30 to 0.50] | 0.45 [0.35 to 0.57] | 0.57 [0.46 to 0.71]
  Day 28: number analyzed (Participants) | 89 | 89 | 0
  Day 28 | 1.10 [0.87 to 1.38] | 0.98 [0.81 to 1.17] |

7. Secondary Outcome: Number of IFNγ Producing Cells/Million PBMCs
Description: IFNγ producing cells as a measurement of cellular immunity will be assessed on a subset (50%) of the participants from each group. IFN-γ Enzyme-Linked ImmunoSpot (Elispot) assay will be performed on isolated peripheral blood mononuclear cells (PBMCs) stimulated with SARS-CoV-2 specific peptides. Data will be reported as number of IFNγ producing cells/million and presented using means and 95% confidence intervals.
Time Frame: Baseline (pre booster), 6, 12 and 18-months post booster vaccination
Reporting Status: Not Posted

8. Secondary Outcome: Frequency of Cytokine-expressing T Cells
Description: Frequency of cytokine-expressing T cells will be assessed on a subset (50%) of participants using Flow cytometry (intracellular staining) on PBMCs samples stimulated with SARS-CoV-2 specific peptides. Data will be reported as frequency (%) of cytokine-expressing T cells presented as means and 95% CI.
Time Frame: Baseline (pre booster), 6, 12 and 18 -months post booster vaccination
Reporting Status: Not Posted

9. Secondary Outcome: Cytokine Concentrations Following PBMCs Stimulation
Description: Cytokine concentrations following PBMCs stimulation will be assessed on a subset (50%) of participants using multiplex cytokine assays. Data will be reported as cytokine concentrations in pg/ml and presented as GMC and 95% CI.
Time Frame: Baseline (pre booster), 6, 12 and 18-months post booster vaccination
Reporting Status: Not Posted

10. Secondary Outcome: Incidence of Unsolicited Adverse Events (AE)
Description: Unsolicited adverse events were collected for 28 days post-booster. Results are reported as the number and percentage of randomised participants in each arm who experienced an unsolicited AE.
Time Frame: 28 days-post booster vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax
Number analyzed (Participants) | 177 | 176
Participants
  Dyspnoea | 3 | 1
  Chest pain | 2 | 1
  Headache | 1 | 0
  Supraventricular tachycardia | 1 | 0
  Acne | 1 | 0
  Mouth ulceration | 1 | 0
  Heavy menstrual bleeding | 0 | 1
  Nasal congestion | 0 | 1
  Administration site pain | 0 | 1
  Road traffic accident | 0 | 2
  Tinnitus | 0 | 1
  No reported AE | 168 | 168

11. Secondary Outcome: Incidence of Medically Attended Adverse Events (AE)
Description: Participants with medically attended AE will be collected for 3 months post booster vaccination. Data will be presented as number of medically attended adverse events. Serious adverse events (SAEs) are reported separately.
Time Frame: 3 months post booster vaccination
Measure: Number; unit: Medically attended adverse events
Groups:
- Controls: Participants who have received three doses of COVID-19 vaccine, with the last dose at least 6 months prior to the study, will be recruited but will not receive any COVID-19 vaccine.
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Controls
Number analyzed (Participants) | 177 | 176 | 143
Medically attended adverse events | 0 | 1 | 0

12. Secondary Outcome: Incidence of Serious Adverse Events (SAE)
Description: Serious adverse events (SAEs) were collected throughout the 24-month follow-up period after booster vaccination. Data are reported as the number of SAEs occurring in each randomised arm.
Time Frame: 24 months post booster vaccination
Measure: Number; unit: Serious adverse events
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Controls
Number analyzed (Participants) | 177 | 176 | 143
Serious adverse events | 5 | 8 | 8

13. Other Pre Specified Outcome: SARS-CoV-2 Infections
Description: SARS-CoV-2 infections were recorded throughout the 24-month follow-up period based on participant self-report of a positive RAT or PCR test. Data are reported as the number of infections occurring in each study arm during this period
Time Frame: 24 months post booster vaccination
Measure: Number; unit: Reported SARS-CoV-2 infections
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Controls
Number analyzed (Participants) | 177 | 176 | 143
Reported SARS-CoV-2 infections | 101 | 85 | 78

ADVERSE EVENTS:
Time Frame: Incidence of Unsolicited Adverse Events (AE) were collected 28 days-post booster vaccination
Arm/Group | Bivalent Moderna (mRNA-1273.214) | Novavax | Controls
All-Cause Mortality (participants affected / at risk) | 0/177 | 0/176 | 0/143
Serious Adverse Events (participants affected / at risk) | 5/177 | 8/176 | 8/143
Other Adverse Events (participants affected / at risk) | 10/177 | 8/176 | 1/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bivalent Moderna (mRNA-1273.214) (N=177) | Novavax (N=176) | Controls (N=143)
Acute pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hand tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infective exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Postpartum sepsis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine rupture (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bivalent Moderna (mRNA-1273.214) (N=177) | Novavax (N=176) | Controls (N=143)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT05658523/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT05658523/SAP_001.pdf